CLINICAL TRIAL: NCT00153192
Title: A Randomized Controlled Clinical Trial of Dronabinol (Marinol) vs Placebo as Add-on Therapy For Patients on Opioids for Chronic Pain
Brief Title: Study to Evaluate the Efficacy of Dronabinol (Marinol) as Add-On Therapy for Patients on Opioids for Chronic Pain
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Sanjeet Narang, Instructor in Anesthesia, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2001-P-000474; BN7894973
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Pain
Keywords: Marinol; Dronabinol; Cannabinoid; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Dronabinol

INTERVENTIONS:
Drug: Marinol (dronabinol)

SUMMARY:
The purpose of this research study is to determine if Marinol alleviates pain in patients with chronic pain who are currently taking opioids.

The study begins with a 2-hour initial visit followed by three 8-hour appointments at Brigham and Women's Hospital. At each 8-hour visit, patients receive a dose of medication and complete surveys relating to pain.

During the first visit a brief examination and a few surveys about pain, quality of life, and medical history are given. The study doctor then determines if the participant continues to qualify for the study.

If qualified for the study, patients receive a daily diary to record pain levels and pain medications; this will take about 5 minutes each day. After completion of the diary, patients begin the 8-hour visits.

Patients visit the Pain Trials Center three times to receive study medication. After taking the study medication, participants remain in the clinic for 8 hours to complete hourly surveys about pain and pain relief.

Subsequent to these visits, patients may enter a 1-month extension where Marinol is taken at home, and pain levels are recorded in a diary. Participants can change the dose of study drug to better control pain and side effects, after speaking with study staff. The study then concludes with a final 30-minute visit to summarize the participant's experience in the clinical trial.

DETAILED DESCRIPTION:
During the informed consent process subjects will be informed that Marinol (Dronabinol) is generally not used for chronic pain and there will be no provision for extended treatment with Dronabinol.

The study comprises two phases, the blinded single-dose phase and the open-label multi-dose phase. There are five visits in all; one baseline visit, three treatment visits in the single-dose phase, and then a final end-of-study visit after the multi-dose phase is over.

Subjects will be initially screened by telephone, and if eligible will present for a baseline visit. This visit will verify enrollment criteria, and will include a history and physical exam, urine pregnancy test if indicated, and baseline assessments. Subjects who meet full enrollment criteria will be randomly allocated to one of the treatment sequences of the single-dose phase.

Single-Dose Phase

The treatment sequence will be a randomized 3-treatment, 3-period crossover trial. Each subject will receive each treatment in a sequence randomly allocated by the Investigational Drug Services Department at Brigham and Women's Hospital. These visits will be scheduled a minimum of 3 days apart, and subjects will be instructed to reschedule if their pain is less than 4/10 on the morning of their visit.

On the days of the treatment visits, subjects will arrive in the Clinical Trials Center at 7-8am, without having taken their morning opioid dose. They will also be fasting, except for clear liquids. They will have a baseline blood sample drawn for level of THC, if any, in their blood. Patients will receive study drug at 8-9 am, and will be monitored for 8 hours, and subsequently discharged home. At the 4- and 8-hour mark, two more blood samples will be drawn. Total amount of blood taken for all three samples together will be less than 10 ml. Subjects who require rescue dosing during the 8-hour study period will take their customary rescue analgesic, be observed in the study center to ensure that they achieve adequate relief of their pain, and then discharged home. A "rescue assessment" will be completed at the time of rescue dosing and will be the final assessment for that treatment session. At the end of the fourth visit (the final treatment visit), prior to discharge, subjects will be offered entry into the one-month open-label extension.

Multi-Dose Phase

Subjects who choose to enter the open-label extension will be provided Marinol tablets which they will then take according to a prearranged titration table. Subjects may titrate upwards for inadequate analgesia or downwards for side effects. Subjects must be on a dose for a minimum of two days prior to upward titration, but may titrate downward at any time due to side effects. Subjects unable to tolerate any regimens will be dropped from the study. Subjects will be required to be on a stable dronabinol regimen during the last week of the study. Subjects who choose to terminate early will be encouraged to present for a termination visit.

Subjects will continue baseline analgesics, including background and rescue opioids as they had been prior to the trial. Downward titration of opioids will be allowed if clinically indicated, per judgment of patient and investigator. Subjects will be contacted weekly at the end of weeks 1, 2, and 3. Data collected during the telephone contacts will relate to pain, medication consumption (study and non-study analgesics), and side effects. Subjects will present for an end-of-study visit at the end of week 4.

ELIGIBILITY:
Inclusion Criteria:

* Chronic somatic nociceptive pain syndromes*, with a minimum pain score on average of 4/10
* Stable doses of opioid analgesics per investigator judgment
* Negative urine pregnancy test in all females with reproductive capacity
* Patients agree to use adequate birth control measures during the study

(*including but not limited to, musculoskeletal pain, neck pain, low back pain, pain due to osteoarthritis, fibromyalgia, failed back surgery syndrome etc.)

Exclusion Criteria:

* Current substance abuse by self-report.
* Chronic pain due to cancer
* Any marijuana use within three months by self-report
* Active litigation, compensation, or disability issues
* Significant baseline nausea, vomiting, sedation, or other symptoms that may compromise the collection of study-related data
* Patients on a baseline opioid regimen that requires opioid dosing more frequently than every 8 hours
* Unstable psychiatric disorders per investigator judgment
* Baseline Beck depression inventory indicating moderate or greater depression, or active suicidality
* Baseline anxiety inventory indicating moderate or greater anxiety
* Patient feels unable to defer morning opioid dose until arrival in the study center
* Patients using Duragesic patch
* Patients receiving opioids via an implanted intrathecal pump

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2001-04; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Single-Dose Phase
- Total pain relief (TOTPAR) at 8 hours
Multi-Dose Phase
- Change in pain score from baseline

SECONDARY OUTCOMES:
Single-Dose Phase
- Sum of pain intensity differences at 8 hours
- Pain and pain relief at all prespecified time points
- SPID for pain bothersomeness at 8 hours
- Side effects scale
- Addiction Research Center Inventory scale of abuse liability
- Patient global assessment at 8 hours
- Changes in mood
- Evoked pain at all prespecified timepoints
- SPID for evoked pain at 8 hours
- Drop outs due to need for rescue analgesia during the 8 hour study phase
- Least squares mean change in pain score by ANCOVA.
- Plasma levels of THC vs. effect of study drug
Multi-Dose Phase
- Time-weighted average of weekly pain assessments collected during study visits and by telephone
- Patient global assessment
- Adverse events
- Quality of life (SF-36) compared to baseline on aggregate score and subscales.
- Sleep scale

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeet Narang, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States